CLINICAL TRIAL: NCT02123069
Title: Sympathetic Nerve Activity and Vascular Function in Women With Uterine Leiomyomata
Brief Title: Vascular Function and Uterine Fibroids
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Joyner, M.D., PI, Mayo Clinic
Other Study IDs: 13-000596
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Leiomyoma
Keywords: Autonomic nervous system; Blood pressure; Blood vessels; Physiological effects of drugs; Vascular stiffness
MeSH Terms: conditions — Leiomyoma | interventions — Acetylcholine; Nitroprusside; Norepinephrine; Phenylephrine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and serum
  No DNA extraction from samples is planned.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with uterine fibroids: * Brachial artery catheter
  * Acetylcholine
  * Nitroprusside
  * Norepinephrine
  * Nitroprusside and phenylephrine
  Interventions: Device: Brachial artery catheter; Drug: Acetylcholine; Drug: Nitroprusside; Drug: Norepinephrine; Drug: Nitroprusside and phenylephrine
- Women without uterine fibroids: * Brachial artery catheter
  * Acetylcholine
  * Nitroprusside
  * Norepinephrine
  * Nitroprusside and phenylephrine
  Interventions: Device: Brachial artery catheter; Drug: Acetylcholine; Drug: Nitroprusside; Drug: Norepinephrine; Drug: Nitroprusside and phenylephrine

INTERVENTIONS:
Device: Brachial artery catheter — A catheter will be placed in the brachial artery by a physician on the study day.
Drug: Acetylcholine — Acetylcholine will be infused into the brachial catheter while blood flow levels in the forearm are measured. Acetylcholine will be infused at the following doses: 1.0, 2.0, 4.0, and 8.0 ug/100 ml tissue/min for 2 minutes each.
Drug: Nitroprusside — Nitroprusside will be infused into the brachial catheter while blood flow levels in the forearm are measured. Nitroprusside will be infused at the following doses: 0.25, 0.5, 1.0, and 2.0 ug/100 ml tissue/min for 2 minutes each.
Drug: Norepinephrine — Norepinephrine will be infused into the brachial catheter while blood flow levels in the forearm are measured. Norepinephrine will be infused at the following doses: 1.0, 2.0, 4.0, and 8.0 ug/100 ml tissue/min for 2 minutes each.
Drug: Nitroprusside and phenylephrine — A single dose of nitroprusside (100 ug) will be infused through an IV; one minute later, a single dose of phenylephrine (150 ug) will be infused.

SUMMARY:
The purpose of this study is to learn how uterine fibroids may be connected to heart disease and high blood pressure. It is not known what causes fibroids, but they frequently occur in women who also have high blood pressure, heart disease, and stroke. The investigators of this study want to learn if certain changes in the blood vessels or nerve activity can put women at risk for these diseases and for fibroids.

DETAILED DESCRIPTION:
The investigators are inviting women, 25-50 years old, who have not gone through menopause to participate in this study. The investigators are looking for some women with uterine fibroids and some without uterine fibroids based on ultrasound or MRI. If the patients have not had a recent ultrasound or MRI of the uterus, a physician can provide one.

Individuals cannot participate if they have high blood pressure, diabetes, or disease in the kidneys, lungs, or blood vessels. Also, individuals who smoke, have high cholesterol, or are obese (BMI is higher than 30) cannot participate. Certain medications, including high blood pressure medications, beta-blockers and anti-depressants, will also limit potential patient participation. The investigators would be happy to review medications for potential participants.

Screen Day:

One of the members of the research team will review the study and the informed consent document with the patient. The patient will have their height, weight, blood pressure, pulse and respirations measured. The patient will also complete three questionnaires. If the patient has not had an ultrasound of the uterus in the last 12 months, a physician will complete one for her.

Study Day:

The patient will need to fast overnight (no eating or drinking). The investigators will draw a blood sample and then do a series of tests on the participant's blood vessels. For some of the tests, medication will be given through an IV. The investigators will also test nerve activity in the nerve on the outer aspect of the leg.

ELIGIBILITY:
Inclusion Criteria:

* Women 25-50 years old
* Premenopausal

Exclusion Criteria:

* Postmenopausal
* Pregnant or currently breastfeeding
* Using blood pressure medications or anti-depression medications
* High blood pressure
* Diabetes
* Disease in the kidneys, lungs, or blood vessels
* Chronic diseases (for example: Crohn's disease, rheumatoid arthritis, bipolar mood disorder, etc.)
* Smoker
* High cholesterol
* BMI higher than 30

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal women, ages 25-50 years old, who have and have not been diagnosed with uterine fibroids. Women will be recruited from Rochester, Minnesota and the surrounding area (including locations in Iowa and Wisconsin). Women eligible to participate will be in good health and not taking medications.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Baseline systolic, diastolic, and mean blood pressures | One day (study day)
Baseline sympathetic nerve activity | One day (study day)
  Nerve "burst" activity will be measured across 10 minutes.

SECONDARY OUTCOMES:
Changes in forearm blood flow levels in response to acetylcholine infusion | One day (study day)
Changes in forearm blood flow levels in response to nitroprusside infusion | One day (study day)
Changes in forearm blood flow levels in response to norepinephrine infusion | One day (study day)
Change in blood pressure in response to infusions of nitroprusside and phenylephrine | One day (study)
  An infusion of nitroprusside will be given, followed by an infusion of phenylephrine one minute later.
Pulse wave velocity (an index of vessel stiffness) | One day (study day)

OTHER OUTCOMES:
Female sex hormone levels | One day (study day)
  Blood samples will be collected to measure levels of estrogen and progesterone.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Joyner, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States